CLINICAL TRIAL: NCT04795323
Title: Proof of Concept (Proof of Intervention Principles) Study Assessing Effects of Technology-Assisted Respiratory Adherence Prototype Version 3 (a Digital Behaviour Change Intervention, DBCI) on Proximal Clinical Outcomes and Mediators (Psychological Mediators, Self-management Behaviours) in Individuals With COPD (IwCOPD)
Brief Title: Proof of Concept Study Assessing Technology-Assisted Respiratory Adherence Prototype Version 3 in Individuals With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0352-2154
Record Dates: First submitted 2021-03-11; First posted 2021-03-12 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: TARA v3.1, only non-pharmacological self-management support (Experimental): Technology-Assisted Respiratory Adherence (TARA) is a digital behaviour change intervention (DBCI) intended to support patients with chronic obstructive pulmonary disease (COPD) in managing their condition by adopting and sustaining clinically recommended (evidence-based) self-management behaviours. TARA was used independently at home by patients via an internet-enabled device and was a fully online digital system that offered guidance on the self-management of COPD, targeting non-pharmacological self-management support (self-monitoring, pursed lip breathing, pacing and energy conservation, and adherence to prescribed rescue medication in TARA version 3.1 (v3.1). The study comprised a screening (pre-TARA) period (which included a 2-week run-in period), a 12-week intervention period (TARA study period), and a follow-up period (post-TARA).
  Interventions: Device: TARA v3.1, only non-pharmacological self-management support
- Cohort 2: TARA v3.2, both non-pharmacological and pharmacological self-management support (Experimental): TARA is a digital behaviour change intervention (DBCI) intended to support patients with COPD in managing their condition by adopting and sustaining clinically recommended (evidence-based) self-management behaviours. TARA is used independently at home by patients via an internet-enabled device and is a fully online digital system that offers guidance on the self-management of COPD, targeting non-pharmacological self-management support (self-monitoring, pursed lip breathing, pacing and energy conservation, and adherence to prescribed rescue medication) in TARA version 3.1 (v3.1). Additionally, in TARA v3.2, pharmacological self-management support module (including modules on inhaler techniques and correct use of inhalers, plus a module to close track inhaler use and symptoms over a 7-day period) was included. The study comprised a screening (pre-TARA) period (included a 2-week run-in period), a 12-week intervention period (TARA study period), and a follow-up period (post-TARA).
  Interventions: Device: TARA v3.2, both non-pharmacological and pharmacological self-management support

INTERVENTIONS:
Device: TARA v3.1, only non-pharmacological self-management support — Technology-Assisted Respiratory Adherence (TARA) is a digital behaviour change intervention (DBCI) intended to support patients with chronic obstructive pulmonary disease (COPD) in managing their condition by adopting and sustaining clinically recommended (evidence-based) self-management behaviours. TARA was used independently at home by patients via an internet-enabled device and was a fully online digital system that offered guidance on the self-management of COPD, targeting non-pharmacological self-management support (self-monitoring, pursed lip breathing, pacing and energy conservation, and adherence to prescribed rescue medication in TARA version 3.1 (v3.1). The study comprised a screening (pre-TARA) period (which included a 2-week run-in period), a 12-week intervention period (TARA study period), and a follow-up period (post-TARA).
  Arms: Cohort 1: TARA v3.1, only non-pharmacological self-management support
Device: TARA v3.2, both non-pharmacological and pharmacological self-management support — Technology-Assisted Respiratory Adherence (TARA) is a digital behaviour change intervention (DBCI) intended to support patients with chronic obstructive pulmonary disease (COPD) in managing their condition by adopting and sustaining clinically recommended (evidence-based) self-management behaviours. TARA was used independently at home by patients via an internet-enabled device and was a fully online digital system that offered guidance on the self-management of COPD, targeting non-pharmacological self-management support (self-monitoring, pursed lip breathing, pacing and energy conservation, and adherence to prescribed rescue medication in TARA version 3.1 (v3.1). The study comprised a screening (pre-TARA) period (which included a 2-week run-in period), a 12-week intervention period (TARA study period), and a follow-up period (post-TARA).
  Arms: Cohort 2: TARA v3.2, both non-pharmacological and pharmacological self-management support

SUMMARY:
The study's primary aim is to assess whether there is a clinically significant reduction in breathlessness in symptomatic individuals with chronic obstructive respiratory disease (IwCOPD) following engagement with Technology-Assisted Respiratory Adherence prototype 3.

The study's secondary aim is to assess whether there is an associated maintenance or increase in activities of daily living to support a positive benefit of Technology-Assisted Respiratory Adherence prototype 3 on breathlessness and whether there is an improvement in the physical activity experience of the patient.

ELIGIBILITY:
Inclusion criteria:

* Individuals with COPD (IwCOPD)
* Male or females
* Age ≥ 40 years
* Current or ex-smokers
* Modified Medical Research Council Dyspnoea Scale (mMRC) score ≥ 2 (i.e. evidence of activity-related breathlessness)
* Patients must have a prescription for either Spiriva Respimat or

Stiolto Respimat as per one of the below scenarios:

1. Participants must have a new prescription for either Spiriva Respimat or Stiolto Respimat (this could include a patient who has never received a maintenance bronchodilator for treatment before, or a patient who was previously on an alternative maintenance bronchodilator who is being switched to Spiriva Respimat or Stiolto Respimat to help with their COPD management).
2. Participants currently on Spiriva Respimat or Stiolto Respimat who could benefit from engagement with Technology-Assisted Respiratory Adherence prototype version 3 (after discussion with their physician).

   * Participants must be on a short-acting bronchodilator ("rescue medication")
   * Participants must be willing to use the study specific activity tracker (Reemo device) and be willing to complete all data collection requirements (within Technology-Assisted Respiratory Adherence prototype version 3) plus on-line questionnaires plus possible phone interview)
   * Fluency in written English
   * Access to a Smartphone with updated browsers installed (or willing to download up-to-date version for the study), and daily home access to internet
   * Need to have personal e-mail account that is used daily

Exclusion criteria:

* Patients with asthma
* Patients with confirmed, suspected or recovered SARS-CoV-2 infection or if the patient had household or other contact with an individual with confirmed SARS-CoV-2 infection.
* Patient with a worsening COPD episode requiring medical intervention within 4 weeks of enrolment
* Patients who have completed a pulmonary rehabilitation (PR) or self-management program in the 3 months prior to enrolment or patients who are currently in a PR program
* Patients prescribed inhaled COPD medications other than Spiriva Respimat plus albuterol or Stiolto Respimat plus albuterol
* Patients with any contraindications for participating in the study (after discussion with their physician).
* Currently enrolled in another investigational device or drug trial, or less than 30 days since ending another investigational device or drug trial(s), or receiving other investigational treatment(s)
* Women who are pregnant, nursing, or who plan to become pregnant while in the study
* Any self-reported medical or neuro-cognitive condition that would limit the ability of the participant to consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Lowcountry Lung and Critical Care, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'.For study data -1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study followed a within-subject pre-post study design and was conducted as a hybrid (clinic visit/remote) study of a software as medical device (SaMD) in individuals with chronic obstructive pulmonary disease (IwCOPD), in a real-world setting.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated if any of the entry criteria were violated.
Groups:
- Cohort 1: TARA v3.1, Only Non-pharmacological Self-management Support: Technology-Assisted Respiratory Adherence (TARA) is a digital behaviour change intervention (DBCI) intended to support patients with chronic obstructive pulmonary disease (COPD) in managing their condition by adopting and sustaining clinically recommended (evidence-based) self-management behaviours. TARA was used independently at home by patients via an internet-enabled device and was a fully online digital system that offered guidance on the self-management of COPD, targeting non-pharmacological self-management support (self-monitoring, pursed lip breathing, pacing and energy conservation, and adherence to prescribed rescue medication) in TARA version 3.1 (v3.1). The study comprised a screening (pre-TARA) period (which included a 2-week run-in period), a 12-week intervention period (TARA study period), and a follow-up period (post-TARA).
- TARA v3.2, Both Non-pharmacological and Pharmacological Self-management Support: Technology-Assisted Respiratory Adherence (TARA) is a digital behaviour change intervention (DBCI) intended to support patients with chronic obstructive pulmonary disease (COPD) in managing their condition by adopting and sustaining clinically recommended (evidence-based) self-management behaviours. TARA was used independently at home by patients via an internet-enabled device and was a fully online digital system that offered guidance on the self-management of COPD, targeting non-pharmacological self-management support (self-monitoring, pursed lip breathing, pacing and energy conservation, and adherence to prescribed rescue medication) in TARA version 3.1 (v3.1). Additionally, in TARA v3.2, pharmacological self-management support module (including modules on inhaler techniques and correct use of inhalers, plus a module to close track inhaler use and symptoms over a 7-day period [medication adherence]) was included. The study comprised a screening (pre-TARA) period (which included a 2-week run-in period), a 12-week intervention period (TARA study period), and a follow-up period (post-TARA).
Period: Overall Study
Arm/Group | Cohort 1: TARA v3.1, Only Non-pharmacological Self-management Support | TARA v3.2, Both Non-pharmacological and Pharmacological Self-management Support
Started (Entered set (ES)) | 4 | 1
Completed | 3 | 1
Not Completed | 1 | 0
Not completed — Did not interact with TARA | 1 | 0

BASELINE CHARACTERISTICS:
Population: Entered set (ES): This subject set includes all enrolled subjects with informed consent who completed the baseline Survey.
Groups:
- Cohort 2: TARA v3.2, Both Non-pharmacological and Pharmacological Self-management Support: Technology-Assisted Respiratory Adherence (TARA) is a digital behaviour change intervention (DBCI) intended to support patients with chronic obstructive pulmonary disease (COPD) in managing their condition by adopting and sustaining clinically recommended (evidence-based) self-management behaviours. TARA is used independently at home by patients via an internet-enabled device and is a fully online digital system that offers guidance on the self-management of COPD, targeting non-pharmacological self-management support (self-monitoring, pursed lip breathing, pacing and energy conservation, and adherence to prescribed rescue medication in TARA version 3.1 (v3.1). Additionally, in TARA v3.2, pharmacological self-management support module (including modules on inhaler techniques and correct use of inhalers, plus a module to close track inhaler use and symptoms over a 7-day period [medication adherence]) was included. The study comprised a screening (pre-TARA) period (which included a 2-week run-in period), a 12-week intervention period (TARA study period), and a follow-up period (post-TARA).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: TARA v3.1, Only Non-pharmacological Self-management Support | Cohort 2: TARA v3.2, Both Non-pharmacological and Pharmacological Self-management Support | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Continuous [Median (Full Range); unit: years] | 71.5 [55 to 79] | NA [NA to NA] — Not shown due to privacy considerations. | 71 [55 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
The Chronic Respiratory - Self Administered Individualized (CRQ-SAI) dyspnea domain score [Median (Full Range); unit: Score on a scale] — The CRQ-SAI questionnaire asks participants to mark important, frequent activities that made them feel out of breath during the last 2 weeks (selected from a list) and they can add additional activity. Participants are then asked to select the most important activities, up to a maximum of 5 activities. For each, the participants will mark their level of shortness of breath; ranging from 1 (worst: "extremely short of breath') to 7 (best: "not at all short of breath"). The CRQ-SAI dyspnea domain score was calculated as the mean of 5 questions, excluding those questions not answered.
  Score on a scale | 2.40 [1.67 to 6.00] | 4.80 [4.80 to 4.80] | 3.00 [1.67 to 6.00]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Chronic Respiratory - Self Administered Individualized (CRQ-SAI) Dyspnea Domain Score at 12 Weeks
Description: The CRQ-SAI questionnaire first asks participants to mark important, frequent activities that made them feel out of breath during the last 2 weeks; they can select these activities from a list, and they can also add additional activities to the list. Participants are then asked to select the most important activities from the list, up to a maximum of 5 activities. Next, for each of these activities, which correspond to questions 1-5, the participants will mark their level of shortness of breath; there are 7 possible answers, ranging from 1 (being the worst: "extremely short of breath') to 7 (being the best: "not at all short of breath"). For each participant, the CRQ-SAI dyspnea domain score was calculated as the mean of numerical answers to the questions 1, 2, 3, 4, 5, excluding those questions not answered. Change was calculated as [score at 12 weeks] - [score at baseline].
Time Frame: Baseline (week 0) and Week 12.
Population: Entered set (ES): This subject set includes all enrolled subjects with informed consent who completed the baseline Survey. Only subjects with post-baseline data are reported.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Cohort 1: TARA v3.1, Only Non-pharmacological Self-management Support | Cohort 2: TARA v3.2, Both Non-pharmacological and Pharmacological Self-management Support
Number analyzed (Participants) | 3 | 1
Score on a scale | 2.00 [0.60 to 4.00] | -0.20 [-0.20 to -0.20]

2. Primary Outcome: Number of Subjects With Increase From Baseline in the CRQ-SAI Dyspnea Domain Score at 12 Weeks of at Least 0.5
Description: Number of subjects with increase from baseline in the CRQ-SAI dyspnea domain score at 12 weeks of at least 0.5, the minimal clinically important difference (MCID). The CRQ-SAI questionnaire first asks participants to mark important, frequent activities that made them feel out of breath during the last 2 weeks. Participants are then asked to select the most important activities from the list, up to a maximum of 5 activities. Next, for each of these activities, which correspond to questions 1-5, the participants will mark their level of shortness of breath; there are 7 possible answers, ranging from 1 (being the worst: "extremely short of breath') to 7 (being the best: "not at all short of breath"). For each participant, the CRQ-SAI dyspnea domain score was calculated as the mean of numerical answers to the questions 1, 2, 3, 4, 5, excluding those questions not answered. Change was calculated as [score at 12 weeks] - [score at baseline].
Time Frame: Baseline (week 0) and Week 12.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: TARA v3.1, Only Non-pharmacological Self-management Support | Cohort 2: TARA v3.2, Both Non-pharmacological and Pharmacological Self-management Support
Number analyzed (Participants) | 3 | 1
Participants | 3 | 0

3. Secondary Outcome: Change From Baseline in Average Number of Steps Measured by the Activity Tracker at Week 12
Description: Daily activity levels were measured using an activity tracker (Reemo) over 2-week periods. The average steps/day were counted over a period of up to 14 days at baseline and at Week 12. A "valid day" was defined as a day where the activity tracker records at least 8 active hours during waking hours (7 am to 10 pm local time for the participant). To calculate the average number of steps/day at baseline (also for Week 12), the data from the prior 14 days were examined. At least 4 valid days out of the 14 days were needed for analysis, but they did not have to be consecutive days. If there were fewer than 4 valid days, the average number of steps/day was not calculated. The average steps/day was calculated as the average over the valid days. Change was calculated as baseline value - week 12 score value.
Time Frame: Baseline (week 0) and Week 12.
Population: as for outcome 1
Measure: Median (Full Range); unit: steps per day
Arm/Group | Cohort 1: TARA v3.1, Only Non-pharmacological Self-management Support | Cohort 2: TARA v3.2, Both Non-pharmacological and Pharmacological Self-management Support
Number analyzed (Participants) | 3 | 1
steps per day | -41.4 [-564.8 to 629.5] | 259.5 [259.5 to 259.5]

4. Secondary Outcome: Change From Baseline in Average Cadence (Steps/Min) Measured by the Activity Tracker at Week 12
Description: Daily activity levels were measured using an activity tracker (Reemo) over 2-week periods. Cadence (steps/min) was calculated as number of steps walked per day divided by the walk time per day (in minutes), then averaged over valid days to produce the average cadence. A "valid day" was defined as a day where the activity tracker records at least 8 active hours during waking hours (7 am to 10 pm local time for the participant). To calculate the average cadence (steps/min) at baseline (also for Week 12), the data from the prior 14 days were examined. At least 4 valid days out of the 14 days were needed for analysis, but they did not have to be consecutive days. If there were fewer than 4 valid days, the average cadence (steps/min) was not calculated. The average cadence (steps/min) was calculated as the average over the valid days. Change was calculated as baseline value - week 12 score value.
Time Frame: Baseline (week 0) and Week 12.
Population: as for outcome 1
Measure: Median (Full Range); unit: Steps per minute
Arm/Group | Cohort 1: TARA v3.1, Only Non-pharmacological Self-management Support | Cohort 2: TARA v3.2, Both Non-pharmacological and Pharmacological Self-management Support
Number analyzed (Participants) | 3 | 1
Steps per minute | 0.00 [-1.63 to 1.19] | 0.67 [0.67 to 0.67]

5. Secondary Outcome: Change From Baseline in the Difficulty Domain of the Clinical Visits PROactive Physical Activity in COPD Instrument (C-PPAC) at Week 12
Description: C-PPAC (with focus on the difficulty domain score). The C-PPAC questionnaire has 12 questions about activities done in the last 7 days, and also records two scores (weekly steps and vector magnitude units) from an activity monitor. Three scores are generated from the C-PPAC (difficulty with physical activity, amount of physical activity and total physical activity). Only the difficulty domain score of the C-PPAC will be analyzed in this study.
  For each participant, the raw score for the C-PPAC difficulty domain is calculated as the sum of the numerical answers to the 10 questions 3-12. Each numerical answer ranges from 0 (most difficult) to 4 (no difficulty). The range of the raw score is 0-40 (with 0 being the most difficult and 40 being no difficulty). This raw score is then scaled to a 0-100 Rasch scaled score (with 0 being the most difficult and 100 being no difficulty). Change was calculated as baseline value - week 12 score value.
Time Frame: Baseline (week 0) and Week 12.
Population: as for outcome 1
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Cohort 1: TARA v3.1, Only Non-pharmacological Self-management Support | Cohort 2: TARA v3.2, Both Non-pharmacological and Pharmacological Self-management Support
Number analyzed (Participants) | 3 | 1
Score on a scale | 14 [-4 to 20] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: After signing the informed consent until the end of study (Week 12), up to 14 weeks.
Description: Entered set (ES): This subject set includes all enrolled subjects with informed consent who completed the baseline Survey.
Arm/Group | Cohort 1: TARA v3.1, Only Non-pharmacological Self-management Support | Cohort 2: TARA v3.2, Both Non-pharmacological and Pharmacological Self-management Support
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 0/4 | 0/1

LIMITATIONS AND CAVEATS:
Due to the small participant population, coupled with a short period of effective availability of TARA for participants in Cohort 1 due to technical issues, the available data were insufficient to draw any conclusions on the efficacy of the software.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT04795323/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT04795323/SAP_001.pdf